CLINICAL TRIAL: NCT02139319
Title: Dose-Escalation of Botulinum Toxin in Subjects With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 43QM1309
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2014-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin (Experimental): Single intra-articular injection
  Interventions: Drug: Botulinum toxin
- Placebo (Placebo Comparator): Single intra-articular injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum toxin
  Arms: Botulinum toxin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of the drug product at each dose level.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee
* Fully weight bearing in the index knee with or without the need for assistive/orthopaedic devices
* Pain score ≥40 mm of the index knee
* Committing to continue using their assistive/orthopaedic device throughout the study using the same regimen

Exclusion Criteria:

* Any infection in the index knee or inflammatory skin disease or other inflammatory diseases at the index knee or the anticipated injection site
* Surgery on the symptomatic knee within the previous 12 months or arthroscopy in the index knee in the past 3 months
* Any painful orthopaedic disorder of the back or hip which is likely to interfere with the safety or efficacy assessments
* A joint disorder other than osteoarthritis in the index knee which could potentially interfere with the safety or efficacy assessments

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Q-Med AB, Study Director — Galderma R&D
Locations (1):
- London, United Kingdom